CLINICAL TRIAL: NCT01914133
Title: Acarbose and Older Adults With Postprandial Hypotension
Acronym: PPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Madden (Other)
Responsible Party: Sponsor-Investigator, Kenneth Madden, Division Head, VGH Division of Geriatric Medicine, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H13-01316; G-13-0001812 (Other Grant/Funding Number: The Heart and Stroke Foundation of Canada (the Foundation))
Record Dates: First submitted 2013-07-22; First posted 2013-08-01 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Other Specified Hypotension; Syncope
Keywords: Acarbose; PPH (Post Prandial Hypotension); Falls; Syncope; Elderly
MeSH Terms: conditions — Syncope | interventions — Acarbose; Glycoside Hydrolase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Postprandial Hypotension (PPH) (No Intervention): Screening Meal Test performed and subject does not meet criteria for Postprandial Hypotension (PPH).
- Placebo (Placebo Comparator): Screening Meal Test performed and subject meets criteria for Postprandial Hypotension (PPH). At second Meal Test subject will receive a placebo and will take a placebo with the first bite of the next 3 meals.
  Interventions: Drug: Placebo
- Acarbose (Active Comparator): Screening Meal Test performed and subject meets criteria for Postprandial Hypotension. During the second Meal Test subject will receive Acarbose 50mg and will take Acarbose 25mg with first bite of each of the next 3 meals.
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Acarbose — Acarbose 50 mg given during Meal Test and Acarbose 25 mg taken with first bite of the next 3 meals.
  Other Names: Glucobay; Precose; Prandase; Alpha-glucosidase inhibitor
  Arms: Acarbose
Drug: Placebo — Placebo given prior to meal the standardized meal
  Other Names: Bayer Material No: 02839265; Acarbose Placebo Tablet
  Arms: Placebo

SUMMARY:
The current proposal will determine if blocking carbohydrate intake in the small intestine with Acarbose can be a possible therapy for older adults with (PPH) Post Prandial Hypotension (a drop of blood pressure after eating), which can result in falls.

DETAILED DESCRIPTION:
Blocking the absorption of carbohydrates at the brush border of the small intestine with acarbose (an alpha-glucosidase inhibitor) seems a promising possibility as a potential therapeutic agent. Although designed as a second-line diabetes drug, this medication has very little risk of hypoglycemia in older adults. In fact the risk of hypoglycemia is extremely low even in patients concurrently taking concurrent hypoglycemia agents (including insulin), and there is almost no risk of hypoglycemia in subjects not on other diabetes medications. Acarbose suppresses postprandial glycemia by slowing small intestinal digestion and absorption of carbohydrate, and has been shown to slow gastric emptying Acarbose has yet to be examined in a prospective fashion in older adults, despite the prevalence of PPH in this patient population. Preliminary, pilot work done in our laboratory on older adults with PPH has demonstrated that the hypotensive response over 90 minutes to a standardized meal was significantly reduced by the administration of acarbose

ELIGIBILITY:
Inclusion Criteria:

* be 65 years of age or older,
* be a non-smoker for at least 5 years
* be referred to the falls clinic at Vancouver General Hospital
* have a Folstein test of cognition > 25/30 to ensure meal log-book compliance

Exclusion Criteria:

* no oral or swallowing issues that would prevent a Meal Test
* subject requiring dialysis due to end-stage renal failure will be excluded
* subjects with evidence on history, physical or blood work of hepatic disease will be excluded since elevated serum transaminases are a potential adverse effect of acarbose
* cannot currently be taking an alpha-glucosidase inhibitor
* cannot have had allergic reactions to alpha-glucosidase inhibitors in the past
* Due to the fact that acarbose is renally excreted, all subjects must have a Creatine Clearance of greater than 25 ml/min
* Subjects with a past history of inflammatory bowel disease, intestinal obstruction, ileus and peptic ulcer disease will be excluded
* Subjects taking carbohydrate-splitting enzymes (such as amylase) will be excluded
* Subjects with chronic respiratory issues requiring treatment will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
The postprandial cardiovascular response to a standardized meal compared between subjects with and without PPH | 2 years
  The postprandial cardiovascular response (mesenteric blood flow, adrenergic response, cerebral blood flow) to a standardized meal will be compared between n=30 subjects with PPH and n= 30 subjects without PPH.

SECONDARY OUTCOMES:
The postprandial glucagon-like peptide-1 (GLP-1) and gastric inhibitory peptide (GIP) response to a standardized meal compared between subjects with and without PPH | 2 years
  The postprandial GLP-1 and GIP response to a standardized meal compared between subjects with and without PPH
The postprandial cardiovascular response between the Acarbose group and the Placebo group will be compared. | 2.5 years
  The postprandial cardiovascular response (mesenteric blood flow, adrenergic response, cerebral blood flow) to a standardized meal between the Acarbose group and the Placebo group will be compared.

OTHER OUTCOMES:
ambulatory blood pressure monitoring (Welch-Allyn, Ambulatory Blood Pressure Monitor(ABPM) 6100S) performed for 24 hours | 1 day
  Starting the day following each meal test, each subject with PPH will take either acarbose 25 mg po tid (prior to each meal) or placebo po tid for one day. During this 24 hour period, each subject will undergo 24 Hr-ABPM (starting at 7 ante meridian (AM) the following day). Each subject will have ambulatory blood pressure monitoring (Welch-Allyn, ABPM 6100S) performed for 24 hours. Each subject will carry a logbook to record time of activity and all meals. Each subject will be given a watch synchronized to the 24-hour blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Madden, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health Research Institute, VGH Research Pavilion Room 186, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madden KM, Feldman B, Meneilly GS. The Effects of Acarbose on the Postprandial Hypotensive Response in Older Adults. Can J Aging. 2025 Sep;44(3):370-376. doi: 10.1017/S0714980825100056. PMID 40719030